CLINICAL TRIAL: NCT05313594
Title: Digital Twin - Modelling Postprandial Triglyceride and Glucose Responses
Status: Completed | Type: Observational
Sponsor: Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Diederik Esser, Clinical Trial Coordinator, Wageningen University and Research
Other Study IDs: NL79685.091.21
Record Dates: First submitted 2022-03-15; First posted 2022-04-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Lipid Metabolism; Glucose Metabolism
Keywords: postprandial; lipids; glucose; dried blood spot; prediction model; metabolic responses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood plasma and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Mixed meal challenge test — Mixed meal consumption followed by postprandial blood sampling
Diagnostic Test: MRI — MRI imaging
Diagnostic Test: DEXA — DEXA scan
Device: Freestyle Libre — Continuous blood glucose measurement
Device: ActivPAL3 — Continuous physical activity measurement

SUMMARY:
Giving personalised dietary advice will help mitigate the postprandial increases in TG and glucose levels, and will assist in the battle against the increase in nutrition-related diseases, such as cardiovascular diseases. Being able to predict postprandial responses, will be a first step to personalised dietary advice.

The primary objective of this study is to validate the prediction model on the effect of a standardized mixed meal challenge on postprandial TG levels in a heterogenous group of middle-aged, overweight to obese individuals. The secondary objectives are 1) to improve the accuracy of the predicted postprandial TG responses by increasing the number of postprandial TG measurements, 2) to determine which parameters can improve the accuracy of the predicted postprandial TG responses, 3) to determine if we can predict the effect of a standardized mixed meal challenge on postprandial glucose levels in a heterogenous group of middle-aged, overweight to obese individuals, and 4) to determine which parameters can improve the accuracy of the predicted postprandial glucose responses. Another objective is to validate dried blood spots postprandial triglyceride concentrations against venous blood concentrations.

There are minor risks for the research subjects of this study. Research subjects will invest approximately 13.5 hours in the study. They will visit the Wageningen University research facility three times and Hospital Gelderse Vallei once.

DETAILED DESCRIPTION:
Elevated triglyceride (TG) and glucose levels are major risk factors for cardiovascular diseases. Therefore, mitigating the postprandial increase in TG and glucose levels may help curb a person's risk of developing cardiovascular diseases. Current strategies to stimulate people to adopt a healthy lifestyle, however, are still insufficient. This is partly due to the fact that nutritional advice is nowadays still given at the population level via general nutrition guidelines, while nutritionist have long been aware that what works for one person may not work for another. Giving personalised dietary advice will help mitigate the postprandial increases in TG and glucose levels, and will assist in the battle against the increase in nutrition-related diseases, such as cardiovascular diseases. Being able to predict postprandial responses, will be a first step to personalised dietary advice.

The primary objective of this study is to validate the prediction model on the effect of a standardized mixed meal challenge on postprandial TG levels in a heterogenous group of middle-aged, overweight to obese individuals. The secondary objectives are 1) to improve the accuracy of the predicted postprandial TG responses by increasing the number of postprandial TG measurements, 2) to determine which parameters can improve the accuracy of the predicted postprandial TG responses, 3) to determine if we can predict the effect of a standardized mixed meal challenge on postprandial glucose levels in a heterogenous group of middle-aged, overweight to obese individuals, and 4) to determine which parameters can improve the accuracy of the predicted postprandial glucose responses. Another objective is to validate dried blood spots postprandial triglyceride concentrations against venous blood concentrations.

Digital twin is an observational study with three visits, including one mixed meal challenge test day.

Study population consists of 38 volunteers, 45-75 year old, BMI between 25-35 kg/m2.

The primary study parameter is the postprandial triglyceride responses in blood upon a mixed meal challenge. The secondary study parameters are: postprandial responses in the blood upon a mixed meal challenge, and extensive phenotyping of the subjects by collecting data on fasting blood profiles of micronutrients, metabolites, and proteins, continuous blood glucose levels (Freestyle Libre), body fat composition (DEXA), liver fat percentage (MRI), habitual dietary intake (FFQ), and physical activity (ActivPAL3).

This study is related to a broad general population. There are minor risks for the research subjects of this study. Consumption of the liquid mixed meal may cause some gastro-intestinal discomfort. Blood sampling will be performed via a cannula and the insertion can be a bit painful and may cause a bruise. The amount of blood that is drawn from subjects is within acceptable limits (total amount collected = 186mL). The radiation dose received during the DEXA scan for measuring body composition, is negligible compared to the average dose each person in the Netherlands receives per year. Research subjects will invest approximately 13.5 hours in the study. They will visit the Wageningen University research facility three times: once for a short screening, once to collect phenotyping data, and once for a mixed-meal challenge test day. In addition, they will visit Hospital Gelderse Vallei once for an MRI measurement.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 45-75 y
* BMI 25-35 kg/m2
* Suitable veins for insertion of cannula

Exclusion Criteria:

* Having a gastro-intestinal disease, such as celiac disease, Crohn's disease, or Ulcerative colitis
* Having a history of intestinal surgery that might interfere with study outcomes, as determined by the medical supervisor. This does not include an appendectomy or cholecystectomy
* Presence of significant systemic diseases, such as diabetes mellitus, cancer, cardiovascular disease or respiratory disease, as determined by the medical supervisor
* Use of medications known to interfere with glucose or lipid homeostasis (e.g. corticosteroids, cholesterol-lowering medication, insulin, metformin), as determined by medical supervisor
* Blood clotting disorders
* Unstable body weight (weight gain or loss >3 kg in the past three months)
* Reported slimming, medically prescribed or other extreme diets
* Alcohol consumption >21 glasses a week
* Anaemia (Hb values <7.5 mmol/L for women and <8.5 mmol/L for men; checked at screening)
* Pregnant, lactating or wishing to become pregnant in the period of the study (self-reported)
* Having a pacemaker, implantable cardioverter-defibrillator, hearing implant, internal insulin pump, neurostimulator, aneurysm clips placed before 1990, or metal splinter in the eye
* Having claustrophobia
* Not willing to give up blood donation during the study
* Food allergies or intolerances for products that we use in the study
* Unwilling to consume non-vegan test meal
* Recent use of antibiotics (<3 months prior to study start)
* Current smokers
* Abuse of soft and/or hard drugs
* Participation in another clinical trial at the same time
* Being an employee of the Food, Health & Consumer Research group of Wageningen Food & Biobased Research or Human Nutrition and Health Department of Wageningen University

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of the study will consist of generally healthy males and females aged 45-75, with a BMI ranging from 25 to 35 kg/m2. For this study, we will include 38 research subjects (aiming at 50% females).
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Postprandial triglycerides blood levels | Baseline
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 15 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 30 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 45 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 60 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 90 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 120 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 150 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 180 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 210 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 240 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 270 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 300 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 330 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 360 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 390 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 420 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 450 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge
Postprandial triglycerides blood levels | 480 minutes post-ingestion
  Postprandial triglyceride responses in blood upon a mixed meal challenge

SECONDARY OUTCOMES:
Postprandial glucose blood levels | Baseline
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 15 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 30 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 45 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 60 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 90 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 120 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 150 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 180 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 210 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 240 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial glucose blood levels | 480 minutes post-ingestion
  Postprandial glucose responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | Baseline
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 15 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 30 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 60 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 90 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 120 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 150 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 180 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 210 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 240 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge
Postprandial insulin blood levels | 480 minutes post-ingestion
  Postprandial insulin responses in blood upon a mixed meal challenge

OTHER OUTCOMES:
Blood glucose profile | Continuous for 5 days
  Continuous blood glucose levels
Physical activity | Continuous for 5 days
  Continuous physical activity levels
Anthropometrics | Baseline
  Waist-to-hip ratio
Body composition | Baseline
  Body composition measurement with Dexa scan
Habitual dietary intake | Baseline
  Habitual dietary intake assessment with FFQ
Liver fat | Baseline
  Liver fat percentage assessment with MRI
Micronutrient levels in blood | Baseline
  Micronutrient levels
Metabolite levels in blood (full profile) | Baseline
  Metabolomics
Protein levels in blood (full profile) | Baseline
  Proteomics
Triglyceride blood levels | Baseline
  Triglyceride measurement in dried blood spots in fingerprick blood upon a mixed meal challenge
Triglyceride blood levels | 120 minutes post-ingestion
  Triglyceride measurement in dried blood spots in fingerprick blood upon a mixed meal challenge
Triglyceride blood levels | 240 minutes post-ingestion
  Triglyceride measurement in dried blood spots in fingerprick blood upon a mixed meal challenge
Triglyceride blood levels | 480 minutes post-ingestion
  Triglyceride measurement in dried blood spots in fingerprick blood upon a mixed meal challenge

CONTACTS AND LOCATIONS:
Overall Officials: Diederik J Esser, PhD, Principal Investigator — Wageningen University & Research
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No